CLINICAL TRIAL: NCT00241202
Title: The Efficacy of the HIV/AIDS Symptom Management Manual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Utah (Other); Massachusetts General Hospital (Other); University of Puerto Rico (Other); Aga Khan University (Other); University of South Africa (Other); Universidad del Turabo (Unknown); Texas A&M University (Other)
Responsible Party: William L. Holzemer, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H642-27289
Record Dates: First submitted 2005-10-13; First posted 2005-10-18 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: HIV; Acquired Immunodeficiency Syndrome
Keywords: signs and symptoms; self care; patient compliance; quality of life
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Signs and Symptoms; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Symptom Management Manual — Participants receive the Symptom Management Manual, and are shown an example. They are given the Manual to take home with them and use.
  Other Names: HIV/AIDS Symptom Management Strategies: A Manual for PLWHA

SUMMARY:
The goals of this research are: 1) To test the efficacy of a self-care symptom management manual by examining whether people who use the manual find it to be useful; 2) To examine symptom and demographic data related to self-care behaviors, symptom control, medication adherence and enhanced quality of life.

The University of California, San Francisco is the coordinating site for this multi-site international study.

DETAILED DESCRIPTION:
People living with HIV/AIDS encounter many psychological, physiological, and cognitive symptoms, such as pain, diarrhea, fever, fatigue, depression, and confusion. These symptoms have been found to restrict a person's daily life significantly. Self-management of multiple HIV and medication side effects symptoms and maintaining optimal quality of life have, therefore, become major daily tasks for people living with HIV/AIDS.

This study is a randomized controlled trial with a two-group repeated measures design to test the efficacy of the symptom management manual. Two groups (experimental and control) will be assessed in a repeated measures design at 3 time points: baseline (time 0), one month (time 1), and two months (time 2). Data will be analyzed using longitudinal mixture modeling.

Comparison(s): HIV-positive patients receiving a symptom management manual and orientation to the manual, compared to HIV-positive patients receiving a nutrition manual and orientation to the manual.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed HIV/AIDS
* Adult (men and women, transgender)
* Presence of at least one symptom within the past week
* Consent
* May or may not be pregnant
* May or may not be on ART
* Able to use the manual with or without family support

Exclusion Criteria:

* Documented diagnosis of dementia
* Unable to understand consent procedure as judged by the person getting consent
* Self-reporting no symptoms within the past week
* Self-reports having had experience with a self-care Symptom Management Manual

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 775 (Actual)
Dates: Start 2005-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Degree of helpfulness (not at all, somewhat, very, extremely) of the symptom management manual at 1 month and 2 months. | 1 month and 2 months

SECONDARY OUTCOMES:
Change in quality of life. | 1 month and 2 months
Change in adherence. | 1 month and 2 months
Change in symptoms. | 1 month and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: William L. Holzemer, RN, PhD, Principal Investigator — University of California, San Francisco
Locations (11):
- United States (7):
  - San Francisco Veteran's Affairs Medical Center, San Francisco, California
  - PositiveHealth Practice, San Francisco, California
  - Jackson Park Hospital, Chicago, Illinois
  - Boston Living Center, Boston, Massachusetts
  - Valley AIDS Clinic - Harlingen, Harlingen, Texas
  - Thomas Street Health Center, Houston, Texas
  - University of Utah Health Science Center, Salt Lake City, Utah
- Nazareth Hospital, Nairobi, Kenya
- Puerto Rico (2):
  - AIDS Clinical Trials Unit, San Juan
  - Casita de Salud Integral Ramón Vicente, Universidad del Turabo, Vega Baja
- PAH ARV Clinic - Tshwane District Hospital, Pretoria, South Africa

REFERENCES:
- See also: Sponsor's website — http://www.aidsnursingucsf.org